CLINICAL TRIAL: NCT05637736
Title: Effects of an Immersive Virtual Reality Intervention Combined With Mindfulness-based Therapy on Mental Health in Nurses During the COVID-19 Pandemic: A Randomized Controlled Trial
Brief Title: Effects of an Immersive Virtual Reality Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nanjing University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Huichao Zhang, Professor, Nanjing University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NUCM22_0708
Record Dates: First submitted 2022-11-24; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Nurse's Role; COVID-19 Pandemic; Mental Stress
MeSH Terms: conditions — COVID-19; Stress, Psychological | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based Stress Reduction by Therapeutic VR (Experimental)
  Interventions: Behavioral: Mindfulness-based Stress Reduction by Therapeutic VR
- mindfulness-based therapy (Active Comparator)
  Interventions: Behavioral: Mindfulness-based Stress Reduction

INTERVENTIONS:
Behavioral: Mindfulness-based Stress Reduction by Therapeutic VR — Therapeutic VR+MBT was provided using a head-mounted display which designed to enclose eyes and block external stimuli almost entirely. Patients can see immersive natural scenes through VR devices and hear stereo sounds through headphones. We uploaded a programme, which was designed to induce recordings of guided meditations (The same as the MBT), musics for meditation and consists of meditation-videos of 40 minutes. We will guide patients to choose their favorite meditation videos, such as forest, seaside, lake, snow mountain, field and so on.
  Arms: Mindfulness-based Stress Reduction by Therapeutic VR
Behavioral: Mindfulness-based Stress Reduction — 39 participates randomized and allocated to this group. MBT was conducted as an 8-week group intervention. Sessions typically began with formal mindfulness meditations that include breathing exercises, prolonged expiratory relaxation, body scan, and meditation. MBT was delivered by the first author, who has specialized training in mindfulness meditation.
  Arms: mindfulness-based therapy

SUMMARY:
Some recent studies demonstrated caregivers may experience negative emotions such as anxiety and sadness, which may also affect normal treatment during the epidemic. As the pandemic continues, mental health support, encouragement , and a sense of purpose are needed to support healthcare workers.

ELIGIBILITY:
Inclusion Criteria:

* Registered nurses (RN) who work in target departments were included. The target departments mainly included internal medicine, surgical, emergency department, where nurses had direct mutual engagement with patients.

Exclusion Criteria:

* Nurses who have not been involved in the COVID-19 volunteer service.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Depression, anxiety, and stress scale (DASS-21) | up to 8 weeks
  The questionnaire of the Chinese version of DASS-21 has a total of 21 items and measures three negative emotional experiences of depression, anxiety and stress
The impact of COVID-19 | up to 8 weeks
  There is a separate questions. "Has COVID-19 affected your mood at work?"(0~10)

CONTACTS AND LOCATIONS:
Locations (1):
- Wu Ye, Nanjing, Jiangsu, China